CLINICAL TRIAL: NCT05493085
Title: Quadratus Lumborum vs Caudal Epidural Block for Perioperative Analgesia in Pediatric Patients Undergoing Upper Abdominal Surgeries.
Brief Title: Quadratus Lumborum vs Caudal Epidural Block for Perioperative Analgesia in Pediatric Patients for Upper Abdominal Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU R 69/2022
Record Dates: First submitted 2022-06-01; First posted 2022-08-09 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Post Operative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum (Active Comparator): Patients will receive Ultrasound-guided quadratus lumborum block
  Interventions: Procedure: Quadratus lumborum block
- Caudal epidural (Active Comparator): Patients will receive single Caudal epidural injection
  Interventions: Procedure: Caudal epidural injection

INTERVENTIONS:
Procedure: Quadratus lumborum block — Ultrasound-guided quadratus lumborum block
  Arms: Quadratus Lumborum
Procedure: Caudal epidural injection — Single Caudal epidural injection
  Arms: Caudal epidural

SUMMARY:
Compare between the analgesic effect of the Ultrasound-guided quadratus lumborum block and single Caudal epidural injection in pediatric patients undergoing surgeries with supraumbilical incisions.

ELIGIBILITY:
Inclusion Criteria:

* Any pediatric patient aged from 2 to 8 years undergoing abdominal Surgery with Supraumbilical umbilical incision

Exclusion Criteria:

* parents refusal to participate in the study,
* previous history of allergy to local anesthetics
* hemodynamic instability
* Coagulopathy,

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Pain score | 24 hours postoperative
  Face, leg, activity, cry and consolability score With score of 0 meaning no pain and requires no intervention and score of 10 indicating the worst imaginable pain requiring rescue analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Wadei, MD, Study Chair — AinShams University, Anesthesia department
Locations (1):
- Ain shams university hospital, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No